CLINICAL TRIAL: NCT00657449
Title: A Double-blind, Double-dummy, Multicenter Randomized Study Of The Efficacy And The Tolerability Of Valdecoxib 40mg Vs Rofecoxib 50mg In The Symptomatic Treatment Of Patients With Ankle Sprain
Brief Title: A Double-blind, Double-dummy, Multicenter, Randomized Study of the Efficacy and Tolerability of Valdecoxib 40 mg Versus Rofecoxib 50 mg in Treating the Symptoms of Ankle Sprain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3471007
Record Dates: First submitted 2008-03-31; First posted 2008-04-14 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Acute Pain
Keywords: sprains and strains
MeSH Terms: conditions — Acute Pain; Sprains and Strains | interventions — valdecoxib; rofecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 2 (Active Comparator)
  Interventions: Drug: rofecoxib

INTERVENTIONS:
Drug: valdecoxib — valdecoxib 80 mg (two 40 mg tablets) by mouth on Day 1 and valdecoxib 40 mg tablet once daily on Days 2-8
  Arms: Arm 1
Drug: rofecoxib — rofecoxib 50 mg (two 25 mg capsules) by mouth once daily for 8 days
  Arms: Arm 2

SUMMARY:
The study compares valdecoxib 40 mg once daily vs. rofecoxib 50 mg one daily in treating the signs and symptoms of acute first- or second-degree ankle sprain. The study also evaluated the disability status, tolerability and safety of these treatments.

DETAILED DESCRIPTION:
A3471007 terminated early (30Sep2004) due to safety concerns about continued usage of rofecoxib after worldwide withdrawal of rofecoxib by Merck & Co Inc

ELIGIBILITY:
Inclusion Criteria:

* Patients had sustained, no more than 48 hours prior to the first dose of study medication, a first- or second-degree ankle sprain of the lateral ligament, specifically: anterior talofibular ligament and/or posterior talofibular ligament and/or calcaneofibular ligament
* At presentation, all patients were to have Patient's Assessment of Ankle Pain Visual Analog Scale (VAS) (0-100mm) of ≥45 mm in the orthostatic position on full weight bearing (ie, moderate to severe pain), had a minimum rating of 2 on the Patient's Global Assessment of Ankle Injury and Patient's Assessment of Normal Function/Activity
* Tthe investigator opinion was that each patient required, and was eligible for, therapy with an anti-inflammatory agent and/or analgesics to control symptoms

Exclusion Criteria:

None reported

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-06-04 (Actual); Primary Completion 2004-10-01 (Actual); Study Completion 2004-10-05 (Actual)

PRIMARY OUTCOMES:
change from baseline in visual analogue scale (VAS) pain intensity | Day 4

SECONDARY OUTCOMES:
patient's assessment of ankle pain VAS (0-100 mm) | Days 1, 4 and 8
patient's and physician's global assessment of ankle injury | Days 1, 4 and 8
patient's and physician's satisfaction assessments | Day 8
patient's assessment of normal function/activity | Days 1, 4 and 8
adverse events, physical examinations, and baseline clinical laboratory values | Adverse Events: Days 1, 4 and 8; Physical examinations: days 1 and 8; Lab tests: day 1

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Brazil (8):
  - Instituto Ortopedico de Goiania, Goiânia, Goiás
  - Centro de Traumatologia e Ortopedia, Goiânia, Goiás
  - Hospital Sao Zacarias, Rio de Janeiro, Rio de Janeiro
  - Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Grupo Hospitalar Conceiçao, Porto Alegre, Rio Grande do Sul
  - Hospital Geral do Grajau, São Paulo, São Paulo
  - Unifesp - Hsp, São Paulo
  - SECONCI, São Paulo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3471007&StudyName=A%20Double-blind%2C%20Double-dummy%2C%20Multicenter%20Randomized%20Study%20Of%20The%20Efficacy%20And%20The%20Tolerability%20Of%20Valdecoxib%2040mg%20Vs%20Rofecoxib%2050mg%20In%20The%20Symptomatic%20Treatment%20Of%20Patients%20With%20Ankle%20Sprain